CLINICAL TRIAL: NCT07149493
Title: Probiotic-containing Nanofiber-based Dental Floss Suppresses Subgingival Red Complex Periopathogens: A Randomized Double-blind Crossover Study
Brief Title: Probiotic Nanofiber Floss and Subgingival Pathogen Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Czech Technology Agency (Unknown); Ministry of Health, Czech Republic (Other Government); RECETOX (Unknown); The University Hospital Brno (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FW02020042
Record Dates: First submitted 2025-08-18; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Dental Hygiene; Probiotics, Periodontitis; Prevention of Dental Caries; Gingivitis and Periodontal Diseases; Periodontal Health; Oral Microbiome
Keywords: probiotics; dental floss; nanofibers; subgingival biofilm; Ligilactobacillus salivarius; red complex; oral microbiome
MeSH Terms: conditions — Periodontitis; Gingivitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking in this study was double-blind. Both participants and investigators were unaware of which type of dental floss-probiotic nanofiber floss or placebo floss-was being used during each phase of the trial. This design was implemented to minimize bias in participant behavior and outcome assessment, ensuring objective evaluation of clinical indices and microbiological results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Floss → Washout → Probiotic Floss (Experimental): Placebo Floss (Invervention 2) → Washout (14 days) → Probiotic Floss (Intervention 1)
  Interventions: Device: Placebo nanofiber floss; Device: Probiotic nanofiber floss
- Probiotic Floss → Washout → Placebo Floss (Experimental): Placebo Floss (Invervention 1) → Washout (14 days) → Probiotic Floss (Intervention 2)
  Interventions: Device: Placebo nanofiber floss; Device: Probiotic nanofiber floss

INTERVENTIONS:
Device: Placebo nanofiber floss — Identical floss without probiotic coating, used under the same conditions.
Device: Probiotic nanofiber floss — Nanofiber floss infused with Ligilactobacillus salivarius (strain BCRC 14759), used twice daily for 14 days.

SUMMARY:
This randomized, double-blind, crossover clinical trial evaluated the effect of a probiotic-containing nanofiber dental floss on subgingival red complex periopathogens and gingival health in periodontally healthy individuals. Thirty male participants underwent two 14-day flossing interventions (probiotic floss and placebo floss), separated by a 14-day washout period. Clinical and microbiological parameters were assessed using standardized indices and multiplex qPCR.

This study was conducted prospectively but is being registered retrospectively to ensure transparency and compliance with NIH guidelines.

DETAILED DESCRIPTION:
The study aimed to validate a targeted subgingival delivery method using Ligilactobacillus salivarius-infused nanofiber floss. Participants received both floss types in a crossover design. Clinical parameters (Approximal Plaque Index and Sulcus Bleeding Index) and microbiological markers (presence of L. salivarius, red complex pathogens, total bacterial DNA) were measured at multiple timepoints. DNA analysis was performed using validated multiplex qPCR protocols. Statistical analysis included non-parametric tests and correlation models. The study was ethically approved and conducted prospectively, but is being registered retrospectively to ensure transparency and support future publication.

Retrospective Registration Note:

This study was originally designed as a method validation investigation to refine subgingival probiotic delivery techniques using a newly developed nanofibre dental floss containing Ligilactobacillus salivarius. At the time of ethics approval and initiation (February 2022), the study was not classified as a clinical trial. However, subsequent interpretation of NIH guidelines suggests that the randomized, blinded, crossover design involving a health-related behavioral intervention meets criteria for interventional clinical research. Accordingly, the investigators now recognize that the study should be registered as a clinical trial. The research team is submitting this retrospective registration to ensure transparency and support future publication. No participant-level outcomes have been modified post hoc, and all data were collected prospectively under full ethical oversight.

ELIGIBILITY:
Inclusion Criteria:

* Male adults (≥18 years) of Czech or Slovak nationality
* ≥20 own teeth
* Good oral hygiene
* Maximum Stage 2 periodontitis

Exclusion Criteria:

* Immunocompromised status
* Systemic illness
* Antibiotic use within 2 months
* Smoking
* Probiotic use during study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Change in Approximal Plaque Index (API) | 14 days of each intervention
  Comparison of clinical indices between pre and post probiotic OR placebo floss periods. Plaque present - 1, not present - 0. Assessment using a probe, one value per tooth.
Change in Sulcus Bleeding Index (SBI) | 14 days of each intervention
  Comparison of clinical indices between pre and post probiotic OR placebo floss periods. Bleeding - 1, not bleeding - 0. Upon probing, one value per tooth.

SECONDARY OUTCOMES:
Detection of L. salivarius DNA in subgingival plaque | 14 days of assigned intervention
  Detection of L. salivarius DNA in subgingival plaque by multiplex qPCR
Quantification of red complex pathogens (P. gingivalis, T. denticola, T. forsythia) | 14 days of assigned intervention
  Quantification of red complex pathogens (P. gingivalis, T. denticola, T. forsythia) with multiplex qPCR
Total bacterial DNA load | 14 days of assigned intervention
  qPCR

CONTACTS AND LOCATIONS:
Locations (1):
- St. Anne's University Hospital, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
Not discussed with the full team

REFERENCES:
- [Derived] Hromcik F, Holochova P, Bohm J, Kuzelova Kostakova E, Pokorny Z, Ruzicka F, Borilova Linhartova P. Probiotic-Containing Nanofiber-Based Dental Floss Suppresses Subgingival Red Complex Periopathogens: A Randomized Double-Blind Crossover Trial. Probiotics Antimicrob Proteins. 2026 Jan 4. doi: 10.1007/s12602-025-10898-4. Online ahead of print. PMID 41484513